CLINICAL TRIAL: NCT00002080
Title: Rifabutin Therapy for the Prevention of Mycobacterium Avium Complex (MAC) Bacteremia in HIV Positive Patients With CD4 Counts = or < 200: Treatment IND Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmacia (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 109A; 087085-999
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-04

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: Rifabutin; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Mycobacterium avium Complex; Bacteremia
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Bacteremia | interventions — Rifabutin

INTERVENTIONS:
Drug: Rifabutin

SUMMARY:
Primary: To provide rifabutin to HIV positive patients in an attempt to prevent or delay Mycobacterium avium Complex (MAC) infection by a daily dose of rifabutin.

Secondary: To further characterize the safety of rifabutin monotherapy in preventing or delaying MAC bacteremia in HIV positive patients with CD4 counts = or < 200.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Any medication with the exception of other investigational drugs not available under a treatment IND, expanded access, or parallel track program.

Patients must have:

* Confirmed HIV infection.
* CD4 cell counts <= 200 cells/mm3.
* No evidence of disseminated MAC disease.
* Informed consent of parent or guardian if 12 to < 18 years of age.

NOTE:

* Pregnant females may be eligible. There are no studies of the safety or efficacy of rifabutin in pregnant women. Rifabutin should be used during pregnancy only if the potential benefit justifies the potential risk to the fetus. In addition, a risk/benefit decision should consider the likelihood of a woman's developing MAC if she does not receive prophylaxis. The risk of developing MAC rises substantially for women with CD4 counts less than 100, although it can also develop in women with higher CD4 counts. Women of reproductive potential who are not pregnant must use contraception. They are encouraged to use means other than oral contraceptives.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Known hypersensitivity to rifabutin, rifampin, or other rifamycins.
* Current infection due to MAC or other mycobacterial disease, or complaints consistent with tuberculosis.

Concurrent Medication:

Excluded:

* Other investigational drugs with the exception of those available under a treatment IND, expanded access, or parallel track program. (Licensed products prescribed for unlabeled indications are not considered investigational.)

Patients with the following prior conditions are excluded:

Prior infection due to MAC or other mycobacterial disease or complaints consistent with tuberculosis.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- PACT, Saint Davids, Pennsylvania, United States

REFERENCES:
- [Background] Gordin F, Masur H. Prophylaxis of Mycobacterium avium complex bacteremia in patients with AIDS. Clin Infect Dis. 1994 Apr;18 Suppl 3:S223-6. doi: 10.1093/clinids/18.supplement_3.s223. PMID 8204774